CLINICAL TRIAL: NCT04345913
Title: A Phase I/II Trial Evaluating the Safety and Efficacy of Eribulin in Combination With Copanlisib in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Testing the Addition of Copanlisib to Eribulin in Metastatic Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-02319; NCI-2020-02319 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 202010089; 10382 (Other: Yale University Cancer Center LAO); 10382 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; copanlisib; eribulin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I (Phase II, eribulin) (Active Comparator): Group I (Phase II): Patients receive eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Eribulin Mesylate; Procedure: Magnetic Resonance Imaging
- Group II (Phase II, DL1, eribulin, copanlisib) (Experimental): Group II (Phase II, DL1): Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Drug: Eribulin Mesylate; Procedure: Magnetic Resonance Imaging
- Phase I, DL1 (eribulin, copanlisib) (Experimental): Phase I, DL1: Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Drug: Eribulin Mesylate; Procedure: Magnetic Resonance Imaging
- Phase I, DL2 (eribulin, copanlisib) (Experimental): Phase I, DL2: Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Drug: Eribulin Mesylate; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
  Arms: Group II (Phase II, DL1, eribulin, copanlisib); Phase I, DL1 (eribulin, copanlisib); Phase I, DL2 (eribulin, copanlisib)
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526 Mesylate; Halaven; Halichondrin B Analog
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase I/II trial studies the side effects and best dose of copanlisib and how well it works when given together with eribulin in treating patients with triple negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as eribulin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving copanlisib and eribulin together may work better in treating advanced stage triple negative breast cancer compared to eribulin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, toxicity profile, dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of copanlisib hydrochloride (copanlisib) in combination with eribulin mesylate (eribulin) in metastatic triple negative breast cancer (TNBC). (Phase I) II. To compare progression free survival (PFS) between eribulin and eribulin plus copanlisib arms in patients with metastatic TNBC treated with prior taxane and anthracycline. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the objective response rate (ORR) and clinical benefit rate (CBR) of the combination. (Phase I) II. To observe and record anti-tumor activity. (Phase I) III. To compare the ORR, CBR (complete response [CR]+partial response [PR]+stable disease [SD] >= 24 weeks) and safety of eribulin and eribulin plus copanlisib arms. (Phase II)

EXPLORATORY OBJECTIVES:

I. To compare PTEN (immunohistochemistry) IHC results between paired baseline tumor biopsy versus at time of disease progression.

II. Assess baseline (pre-treatment) tumor tissue mutation or gene expression profiles to correlate treatment response.

III. Assess intrinsic and adaptive resistance mechanisms by analyzing pre and post treatment biopsies for gene expression and proteomic changes.

IV. Determine circulating tumor DNA (ctDNA) mutation profiles at baseline and changes in mutation profile and variant allele frequencies (VAFs) on cycle 2 day 1 (C2D1) and at disease progression compared to baseline to correlate with treatment response.

V. Assess circulating biomarkers predictive of treatment response. VI. Assess plasma and serum proteomics and metabolomics predictive of treatment response.

VII. To compare the ORR, CBR, PFS of eribulin and eribulin plus copanlisib arms in patients with tumors harboring mutations in PIK3CA/ PTEN or with loss of PTEN expression by IHC on baseline tumor biopsy.

VIII. To compare the ORR, CBR, PFS of eribulin and eribulin plus copanlisib arms in patients with tumors lacking PIK3CA/ PTEN pathway alterations.

IX. To compare the ORR, CBR, PFS of eribulin and eribulin plus copanlisib arms in patients with tumors harboring loss of PTEN expression by IHC in pre-treatment metastatic site (in patients with available tissue from metastatic site).

X. To compare PTEN IHC results between paired archival primary tumor versus (vs.) baseline tumor biopsies.

XI. To assess targeted inhibition by copanlisib and eribulin by measuring treatment induced changes in phosphorylated (phospho)-AKT (T308), phospho-AKT (S473), phospho-histone H3, and inhibition of apoptosis (cleaved caspase 3) between post-treatment tumor (C2D1-2) versus baseline.

XII. To compare the ORR, CBR, PFS of eribulin and eribulin plus copanlisib arms in patients with tumors harboring mutations in PIK3CA/PTEN by circulating tumor deoxyribonucleic acid (ctDNA) at baseline, and potential changes over time.

OUTLINE: This is a phase I dose-escalation study of copanlisib and eribulin followed by a phase II study. Patients are randomized to 1 of 2 groups.

Phase I, DL1: Patients receive copanlisib (45 mg) intravenously (IV) over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Phase I, DL2: Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Group I (Phase II, eribulin): Patients receive eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Group II (Phase II, eribulin + copanlisib, DL1): Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo a computed tomography (CT) scan and/or magnetic resonance imaging (MRI) at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.

After completion of study treatment, patients are followed every 3 months for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients must have metastatic or unresectable carcinoma of the breast that is estrogen receptor (ER) negative (less than 10%), progesterone receptor (PR) negative (less than 10%), and HER2 negative/unamplified
* Patients must have had prior treatment with an anthracycline and taxane in the neoadjuvant, adjuvant, or metastatic setting, unless contraindicated or deemed to be suboptimal therapy per the treating physician
* Patients must have progressed on at least one and not more than five prior chemotherapy regimens, including in the neoadjuvant, adjuvant, and metastatic settings. Prior chemotherapy in the neoadjuvant and/or adjuvant setting counts as one prior line. Prior endocrine therapy, anti-HER2 directed therapies, PARP inhibitors, immunotherapy alone, or other targeted therapy will not count as a prior therapy line, as long as the patient meets the eligibility criteria prior to enrollment. Immunotherapy combined with chemotherapy will be considered one line
* All patients must agree to provide archival tumor material (most recent archival tumor tissue immediately prior to enrollment is strongly preferred) for research and must agree to undergo research tumor biopsy before treatment if presence of easily accessible lesions (judged by the treating physician). For patients with bone only disease, or patients without easily accessible lesions for the baseline research biopsy, availability of archival tumor material (2 x 4-5 micron section unstained slides, plus 15-20 x 10 micron section unstained slides or a tumor rich block) from previous breast cancer diagnosis or treatment is required for PTEN and PIK3CA analysis
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of copanlisib in combination with eribulin in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (=< 3 x institutional ULN for patients with Gilbert syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Lipase =< 1.5 x ULN
* Creatinine < 1.5 mg/dL AND glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2
* International normalized ratio (INR) =< 1.5 x ULN
* Partial thromboplastin time (PTT) =< 1.5 x ULN
* Patients with history of known type I or type II diabetes must have a fasting glucose level of < 120 mg/dL on at least 2 separate occasions or glycosylated hemoglobin measurement (HbA1c) < 8.5% at screening within 14 days prior to registration
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and INR/PTT is stable
* Prophylactic antiemetics may be administered according to standard practice. The routine use of standard antiemetics, including 5-HT3 blockers, such as granisetron, ondansetron, or an equivalent agent, is allowed as needed, as long as corrected QT (QTc) interval on baseline electrocardiogram (ECG) < 480 msec. The use of corticosteroids as antiemetics prior to copanlisib administration will not be allowed
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial provided they are on a stable regimen of anti-retroviral therapy (ART) with no medications otherwise prohibited by this protocol (e.g. drug-drug interactions)
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. For patients with history of treated brain metastases, brain scans will be performed within 6 weeks of study enrollment. During study enrollment in the phase 2 portion of the study, brain MRI will be performed every 12 weeks or sooner if clinically-indicated in all patients with history of known brain metastases
* For phase 1 portion of the study only: patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy. This is not allowed for phase 2 portion of the study
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. Patients with history of known congestive heart failure (left ventricular ejection fraction [LVEF] < 50%) must have documented LVEF >= 50% within 12 months of study enrollment
* Known mutation status for PIK3CA and PTEN from archival tumor tissue analysis
* The effects of copanlisib on the developing human fetus are unknown. For this reason and because maternal toxicity, developmental toxicity and teratogenic effects have been observed in nonclinical studies and PI3K inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 1 month after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3.5 months after completion of study treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks of treatment start (cycle 1 day 1 [C1D1])
* Patients who have had prior treatment with nitrosoureas or mitomycin C
* Patients who have had prior treatment with eribulin
* Patients who have had prior treatment with PI3K/mTOR/AKT pathway inhibitor
* Clinically significant ECG abnormality, including prolonged corrected QT (QTc) interval > 480 msec or history of risk factors for Torsades de Pointes (TdP) (i.e. congestive heart failure, hypokalemia, hypomagnesemia, bradyarrhythmias, family history of long QT syndrome)
* Patients with pre-existing neuropathy of grade 2 or higher
* Myeloid growth factors within 7 days prior to treatment start
* Platelet transfusion within 7 days prior to treatment start
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Immunosuppressive therapy is not allowed while on study
* Known tumor AKT mutation from archival tumor tissue analysis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, PI3K inhibitors, or other agents used in study
* Copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from 14 days prior to enrollment until the end of the study. Other medications that are prohibited while on copanlisib treatment:

  * Herbal medications/preparations (except for vitamins)
  * Anti-arrhythmic therapy other than beta blockers or digoxin
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the CT/MRI screening. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening. Patients may be using topical or inhaled corticosteroids. Short-term (up to 7 days) systemic corticosteroids above 15 mg prednisolone or equivalent will be allowed for the management of acute conditions (e.g., treatment non-infectious pneumonitis). The use of corticosteroids as antiemetics prior to copanlisib administration will not be allowed
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients with non-healing wound, ulcer, or bone fracture. Patients with compression or pathologic fractures that are stable in the opinion of the investigator may be enrolled, as long as the bone fracture is not felt to pose a high likelihood of treatment delay or difficulties in treatment adherence as per the judgement of the investigator
* Patients with active, clinically serious infections > grade 2 (Common Terminology Criteria for Adverse Events Version 5.0 [CTCAEv5.0]) (viral, bacterial or fungal infection)
* History of known Pneumocystis jiroveci pneumonia (PJP) infection
* Patients with arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Concurrent diagnosis of pheochromocytoma due to risk of hypertension with copanlisib
* Uncontrolled hypertension (defined as blood pressure >= 150/90 mm/Hg) despite optimal medical management (per investigator's opinion)
* Proteinuria as estimated by urine protein/creatinine ratio > 3.5 g/g on random urine sample or grade >= 3 as assessed by 24-hour urine protein collection
* Patients with history of or current uncontrolled autoimmune disease. Patients who have adrenal or pituitary insufficiency who are stable on replacement therapy (i.e. thyroxine or physiologic corticosteroid replacement therapy that meets concomitant medication restrictions) are allowed. Limited exceptions may be made to this after discussion with the study principal investigator (PI)
* Patients with congenital QT prolongation
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Pregnant women are excluded from this study because copanlisib is a PI3K inhibitor agent and eribulin is an anti-tubulin agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with copanlisib and eribulin, breastfeeding should be discontinued if the mother is treated with copanlisib and/or eribulin. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2026-05-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nusayba Bagegni, Principal Investigator — Washington University School of Medicine
Locations (43):
- United States (43):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 patients received study treatment (8 patients in Phase I and 16 patients in Phase II). There were 9 additional patients that signed consent and were never treated. This includes 6 screen fails and 3 patients that were not treated and withdrawn prior to receiving study therapy.
Period: Overall Study
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib) | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib)
Started | 6 | 2 | 8 | 8
Completed | 6 | 2 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib) | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib) | Total
Number analyzed (Participants) | 6 | 2 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 6 | 8 | 21
  >=65 years | 1 | 0 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.33 (11.02) | 42.5 (23.33) | 58.00 (7.73) | 50.13 (6.22) | 52.17 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8 | 8 | 24
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 1 | 8 | 7 | 20
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 5 | 3 | 9
  White | 3 | 1 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8 | 8 | 24
Eastern Cooperative Oncology Score (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status Scale (0-5) is a standard criteria for measuring how disease impacts a patient's daily living abilities or performance status.
  0, fully active, can carry out pre-disease performance without restriction
  1. restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. ambulatory and capable of all selfcare but unable to carry out any work activities
  3. capable of only limited selfcare; confined to bed or chair over 50% of waking hours
  4. completely disabled; cannot carry on any selfcare
  5. dead
  Participants
    ECOG 0 | 2 | 0 | 6 | 2 | 10
    ECOG 1 | 4 | 2 | 2 | 6 | 14
PTEN/PIK3CA Mutation [Count of Participants; unit: Participants]
  No Mutation | 4 | 2 | 6 | 7 | 19
  Yes Mutation | 2 | 0 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Eribulin (MTD) (Phase I)
Description: MTD is defined as the highest dose level of eribulin at which at most 1 of 6 patients experience a dose limiting toxicity during the observation window.
Time Frame: Up to 28 days
Population: 6 patients in DL1 and 2 patients in DL2.
Measure: Number; unit: mg/m^2
Groups:
- Phase I, DL and DL2 (Eribulin, Copanlisib): Phase I, DL1 and DL2: DL1 patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. DL2 patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles for both dose levels repeat every 21 days in the absence off disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
Arm/Group | Phase I, DL and DL2 (Eribulin, Copanlisib)
Number analyzed (Participants) | 8
mg/m^2 | 1.1

2. Primary Outcome: Recommended Phase 2 Dose of Eribulin (RP2D) (Phase I)
Description: RP2D is the maximum tolerated dose of eribulin at which at most 1 of 6 patients experience a dose limiting toxicity during the observation window.
Time Frame: Up to 28 days
Population: 6 patients in DL1 and 2 patients in DL2
Measure: Number; unit: mg/m^2
Groups:
- Phase I, DL1 (Eribulin, Copanlisib): Phase I, DL1 and DL2: DL1 patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. DL2 patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.4 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles for both dose levels repeat every 21 days in the absence off disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib)
Number analyzed (Participants) | 8
mg/m^2 | 1.1

3. Primary Outcome: Maximum Tolerated Dose of Copanlisib (MTD) (Phase I)
Description: MTD is defined as the highest dose level of copanlisib at which at most 1 of 6 patients experience a dose limiting toxicity during the observation window.
Time Frame: Up to 28 days
Population: 6 patients in DL1 and 2 patients in DL2
Measure: Number; unit: mg
Arm/Group | Phase I, DL and DL2 (Eribulin, Copanlisib)
Number analyzed (Participants) | 8
mg | 45

4. Primary Outcome: Recommended Phase 2 Dose of Copanlisib (RP2D) (Phase I)
Description: RP2D is the maximum tolerated dose of copanlisib at which at most 1 of 6 patients experience a dose limiting toxicity during the observation window.
Time Frame: Up to 28 days
Population: 6 patients in DL1 and 2 patients in DL2
Measure: Number; unit: mg
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib)
Number analyzed (Participants) | 8
mg | 45

5. Primary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of measurable target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions. Patients who have not experienced progression or death will be censored at last follow up. PFS will be estimated using the Kaplan-Meier product limit estimator.
Time Frame: From date of treatment start to date of progression or death, assessed up to 36 months
Population: Phase II patients only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib)
Number analyzed (Participants) | 8 | 8
months | 3.9 [0.4 to NA] — When fewer than half of participants have experienced disease progression, the median PFS and its upper CI bound may not be estimable. Even when the median is reached, the upper bound can still be NE (NA) if there are too few events beyond that point. | 3.3 [1.7 to 5.4]
Statistical Analysis 1: Comparison: Group I (Phase II, Eribulin) vs Group II (Phase II, DL1, Eribulin, Copanlisib); Test type: Other — This test is used to compare the survival distributions of different groups in a survival analysis. It's a nonparametric test; p = 0.5259, Log Rank

6. Secondary Outcome: Objective Response Rate (ORR) (Phase I)
Description: ORR is defined as the proportion of patients with complete response, partial response by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Per RECIST 1.1, target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Population: Phase I patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib)
Number analyzed (Participants) | 6 | 2
Participants | 0 | 1

7. Secondary Outcome: Clinical Benefit Rate (CBR) (Phase I)
Description: CBR defined as the proportion of patients with clinical benefit (complete response, partial response and stable disease lasting > 24 weeks) per RECIST v1.1 in the overall population, and by PTEN/PIK3CA mutation status based on archival tumor tissue next generation sequencing. Per RECIST 1.1, target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither 30% shrinkage of longest diameter of target lesions to qualify for PR nor 20% increase in longest diameter of target lesion to qualify for PD, for a period of time greater than 24 weeks.
Time Frame: Up to 36 months
Population: Phase I patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib)
Number analyzed (Participants) | 6 | 2
Participants | 0 | 1

8. Secondary Outcome: ORR (Phase II)
Description: as for outcome 6
Time Frame: Up to 36 months
Population: Phase II patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib)
Number analyzed (Participants) | 8 | 8
Participants | 0 | 2

9. Secondary Outcome: CBR (Phase II)
Description: CBR is defined as the proportion of patients with clinical benefit (complete response, partial response, and stable disease lasting ≥ 24 weeks) per RECIST v1.1 in each arm. Per RECIST 1.1, target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither 30% shrinkage of longest diameter of target lesions to qualify for PR nor 20% increase in longest diameter of target lesion to qualify for PD, for a period of time greater than 24 weeks.
Time Frame: Up to 36 months
Population: Phase II patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib)
Number analyzed (Participants) | 8 | 8
Participants | 0 | 3

10. Secondary Outcome: PFS (Phase I)
Description: PFS is defined from date of treatment start to date of progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of measurable target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions. Patients who have not experienced progression or death will be censored at last follow up. PFS will be estimated using the Kaplan-Meier product limit estimator.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 36 months
Population: Phase I patients only
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I, DL1 (Eribulin,Copanlisib): Phase I, DL1: Patients receive copanlisib (45 mg) IV over 1 hour and eribulin (1.1 mg/m^2) IV over 2 to 5 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT scan and/or MRI at screening, cycle 3 day 1, and every 9 weeks thereafter. Patients also undergo a biopsy at baseline, cycle 2 day 1, and at time of disease progression as well as blood sample collection at baseline, cycle 2 day 1, every 9 weeks and at time of disease progression.
Arm/Group | Phase I, DL1 (Eribulin,Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib)
Number analyzed (Participants) | 6 | 2
months | 2.3 [1.2 to NA] — When fewer than half of participants have experienced disease progression, the median PFS and its upper CI bound may not be estimable. Even when the median is reached, the upper bound can still be NE (NA) if there are too few events beyond that point. | 2.6 [2.0 to NA] — When fewer than half of participants have experienced disease progression, the median PFS and its upper CI bound may not be estimable. Even when the median is reached, the upper bound can still be NE (NA) if there are too few events beyond that point.
Statistical Analysis 1: Comparison: Phase I, DL1 (Eribulin,Copanlisib) vs Phase I, DL2 (Eribulin, Copanlisib); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.7060, Log Rank

11. Other Pre Specified Outcome: Tumor Tissue Mutation or Gene Expression Profiles
Description: Will correlate with treatment response
Time Frame: Up to 36 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Intrinsic and Adaptive Resistance Mechanisms
Description: Will analyze pre and post treatment biopsies for gene expression and proteomic changes.
Time Frame: Baseline up to 36 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: ctDNA Mutation Profiles and Changes in Mutation Profile and Variant Allele Frequencies (VAFs)
Description: Will determine ctDNA mutation profiles at baseline and changes in mutation profile and VAFs on C2D1 and at disease progression compared to baseline to correlate with treatment response.
Time Frame: Baseline, cycle 2 day 1 (C2D2), and at disease progression
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Circulating Biomarkers Predictive of Treatment Response
Time Frame: Up to 36 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Plasma and Serum Proteomics and Metabolomics Predictive of Treatment Response
Time Frame: Up to 36 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: PTEN IHC Results
Description: Will compare PTEN IHC results at disease progression compared to baseline.
Time Frame: Up to 36 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: PFS
Description: PFS is defined from date of treatment start to date of progression or death. Patients who have not experienced progression or death will be censored at last follow up. Measured by treatment arm in patients with TNBC harboring mutations in PIK3CA/ PTEN or loss of PTEN expression by IHC of baseline (pre-treatment) biopsy and by treatment arm in patients with TNBC harboring mutations in PIK3CA/ PTEN by ctDNA at baseline (pre-treatment) biopsy and potential changes over time. PFS will be estimated using the Kaplan-Meier product limit estimator.
Time Frame: From date of treatment start to date of progression or death, assessed up to 36 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Target Inhibition of PI3K Pathway and Mitotic Arrest
Description: Using phospho-AKT and phospho-histone H3 with eribulin plus copanlisib versus eribulin alone.
Time Frame: Up to 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from start of treatment through follow up. Patients removed due to unacceptable AE(s), were followed until resolution or stabilization of the AE. Median AE length of follow-up was 62.5 days (full range 7-244 days). All-cause mortality was collected from start of treatment through completion of follow-up. Overall median length of follow-up was 268 days (full range 7-771 days).
Arm/Group | Phase I, DL1 (Eribulin, Copanlisib) | Phase I, DL2 (Eribulin, Copanlisib) | Group I (Phase II, Eribulin) | Group II (Phase II, DL1, Eribulin, Copanlisib)
All-Cause Mortality (participants affected / at risk) | 4/6 | 2/2 | 5/8 | 8/8
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/2 | 1/8 | 5/8
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, DL1 (Eribulin, Copanlisib) (N=6) | Phase I, DL2 (Eribulin, Copanlisib) (N=2) | Group I (Phase II, Eribulin) (N=8) | Group II (Phase II, DL1, Eribulin, Copanlisib) (N=8)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Rhinovirus (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Acute renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, DL1 (Eribulin, Copanlisib) (N=6) | Phase I, DL2 (Eribulin, Copanlisib) (N=2) | Group I (Phase II, Eribulin) (N=8) | Group II (Phase II, DL1, Eribulin, Copanlisib) (N=8)
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 6
Eosiniphilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Fluid in ears (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Periorbital edema (Eye disorders) | 1 | 0 | 0 | 0
itching/discharge from R eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hemorrhoidal hemorhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Axillary lymphadenopathy (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 0 | 4 | 5
Fever (General disorders) | 0 | 0 | 0 | 2
Flu-like symptoms (General disorders) | 1 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 2
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 1
Shingles (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gluted cleft injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 4
BUN increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Cardiac troponin T increased (Investigations) | 1 | 0 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0 | 0
Creatinine decreased (Investigations) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 1 | 0 | 0
BUN decrease (Investigations) | 0 | 0 | 0 | 1
Elevated blood protein (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 1 | 2 | 4
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 2 | 3 | 5
Platelet count decreased (Investigations) | 1 | 0 | 0 | 2
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 1 | 1 | 1 | 0
White blood cell decreased (Investigations) | 4 | 1 | 4 | 7
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0 | 5 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Firm nodal mass in right supraclavicular region (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphadenopathy in lower left cervical chain and left supraclavicular region (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 5
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Intermittant itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Radiation fibrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 3
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04345913/Prot_SAP_000.pdf
  • Informed Consent Form: Research Study Informed Consent Document - Phase 1 (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04345913/ICF_001.pdf
  • Informed Consent Form: Research Study Informed Consent Document -Phase 2 (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04345913/ICF_002.pdf